CLINICAL TRIAL: NCT03206268
Title: Correlation in Retinal Nerve Fiber Layer Thickness in Uveitis and Healthy Eyes Using Scanning Laser Polarimetry and Optical Coherence Tomography
Brief Title: RNFL Thickness Measurements Obtained Using SD-OCT and SLP Using GDx Variable Corneal Compensation
Acronym: Real
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0303
Record Dates: First submitted 2017-04-21; First posted 2017-07-02 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2017-04

CONDITIONS: Uveitis
Keywords: retinal nerve fiber layer thickness; uveitis; SD-OCT; GDx VCC
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy eyes
  Interventions: Device: SD-OCT and SLP using GDx variable corneal compensation
- uveitis eyes
  Interventions: Device: SD-OCT and SLP using GDx variable corneal compensation

INTERVENTIONS:
Device: SD-OCT and SLP using GDx variable corneal compensation — RNFL thickness measurements obtained using SD-OCT and SLP using GDx variable corneal compensation

SUMMARY:
The aim of this study is to evaluate the correlation of retinal nerve fiber layer (RNFL) thickness measured using spectral domain optical coherence tomography (SD-OCT) and scanning laser polarimetry (SLP) in uveitic eyes compared to healthy eyes.

A descriptive, observational, prospective, consecutive, cross-sectional, controlled, mono-center case series was conducted from May to October 2015. Clinical characteristics, best-corrected visual acuity, intra-ocular pressure, RNFL thickness measurement with SD-OCT and SLP using GDx variable corneal compensation (GDx VCC) were performed for each patient. An evaluation of anterior chamber inflammation with laser flare cell meter was also carried out. Correlations between SD-OCT and GDx VCC RNFL measurement were evaluated by linear regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years,
* best-corrected visual acuity better than or equal to 20/40,
* spherical refraction between -6.00 and +3.00 diopters,
* no retinal disease or non-glaucomatous neuropathy, and no ophthalmic surgery in the past 6 months.

Exclusion Criteria:

* Healthy eye were excluded in case of consecutive and reliable abnormal standard automated perimetry with abnormal Glaucoma Hemifield Test and pattern standard deviation outside 95% of normal limits, and optic nerve damage (asymmetric cup-to-disc ratio ≥ 0.2, rim thinning, notching, excavation, or retinal nerve fiber layer defect).
* any history of ophthalmic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sixty-eight consecutive patients were screened between May 2015 and October 2015, 3 (4.4%) of whom were excluded based on poor OCT quality criteria, 7 (10.3%) for poor GDx VCC quality criteria, and 4 (5.9%) for poor visual field quality or reliability criteria. Fifty-four patients were included and divided into two groups: 50 healthy eyes in 29 patients and 42 uveitic eyes in 25 patients. Of these 42-uveitic eyes, 25 eyes (59.5%) had active uveitis and 17 eyes (40.5%) had inactive uveitis
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2015-10-31 (Actual); Study Completion 2015-10-31 (Actual)

PRIMARY OUTCOMES:
Retinal nerve fiber thickness (RNFL) | at inclusion
  measures are made with spectral domain optical coherence tomography (SD-OCT) in micrometer
Retinal nerve fiber thickness (RNFL) | at inclusion
  measures are made with scanning laser polarimetry (SLP) in micrometer

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Denis, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Croix-Rousse University Hospital, Lyon, France